CLINICAL TRIAL: NCT00252577
Title: Genetic Studies of Psychiatric Illness
Brief Title: Genetic Predictors of Lithium Response in Bipolar Disorder
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: MHBA-023-05S
Record Dates: First submitted 2005-11-09; First posted 2005-11-11 (Estimated); Results first posted 2020-01-29 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Bipolar Disorder
Keywords: Lithium; Pharmacogenetics
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA from patients with bipolar disorder
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Group 1: Veterans with bipolar disorder
  Interventions: Drug: Lithium treatment

INTERVENTIONS:
Drug: Lithium treatment — Lithium is a standard treatment for bipolar disorder. Patients will be stabilized on lithium monotherapy over a 3 month period, observed for one month, and then followed every 2 months in maintenance phase for 2 years

SUMMARY:
The purpose of this study is to identify genetic predictors of lithium response in bipolar disorder.

DETAILED DESCRIPTION:
The long term focus of this research program has been identification of genes for bipolar disorder. The investigators have recently obtained evidence from several lines of investigation to support the role of the gene for G protein receptor Kinase 3(GRK3) in bipolar disorder. Work to replicate and extend these results is continuing under NIH funding. In this clinical the investigators will extend the investigators' work into Pharmacogenetics to attempt to identify genes that are associated with medication response in bipolar disorder. Lithium is the first mood stabilizer medication and remains a mainstay of treatment. Many patients have an excellent response to lithium, tolerate it well, and are stabilized for years, while others do not. The reasons for this difference in response are unclear, but it is likely that genetic factors make a substantial contribution. The lack of good predictors of response frequently result in a time consuming trial and error clinical process to find the best medication. Such a trial and error process can take months with prolongation of patient suffering. Hence, there is a strong clinical need for predictors. The investigators have conducted a preliminary study with 92 lithium responders and 92 non-responders identified through retrospective detailed history and chart review. These subjects have been genotyped at 88 single nucleotide polymorphism (SNP) markers in 9 candidates genes relevant to lithium presumed mechanism of action for bipolar disorder. Four SNP markers in three genes showed nominally significant association to lithium response. One of the SNPs in the gene for neurotrophic receptor tyrosine kinase 2 (NTRK2), the receptor for brain-derived neurotrophic factor (BDNF), showed a strong association in patients who had predominantly euphoric a opposed to dysphoric mania (p=0.0005). Many data argue for the role of BDNF in the mechanism of antidepressants and mood stabilized action as well as susceptibility to bipolar disorder. No association was observed in those with dysphoric mania. This suggests that variations in this gene may operate in a clinically and genetically distinct subset of patients. It also argues for the importance of incorporating clinical subtypes into such analyses. These pilot results are preliminary but suggest the feasibility of such an approach. The investigators will conduct a prospective trial of lithium monotherapy in 100 patients with bipolar disorder. 200 patients who are unstable, mildly to moderately ill and not on lithium will be screened and then entered into 16-week stabilization phase where they will be treated and switched to lithium monotherapy. Patient stable on lithium will also be entered and other mediations withdrawn. After stabilization patients will be followed for one year or until a mood episode requires intervention. It is expected that 50% of patients will be stabilized and therefore 100 patients will enter the maintenance phase. Time to relapse and pharmacological intervention will be the primary outcome measure. This prospective sample will be used to replicate previous results at the NTRK2 and other genes. Analyses will be conducted to test for differences in survival curves between different genotypic group. Genomic control methods will be employed to detect or correct for possible stratification and heterogeneity. Clinical features of illness such as dysphoric mania, family history and rapid cycling will be employed as co-variates. Multivariate methods will also be employed in order to attempt to develop a multi-gene predictor of lithium response.

ELIGIBILITY:
Inclusion Criteria:

* Are 18 years of age or older;
* Have a diagnosis of Bipolar Affective Disorder, I or II;
* Have no contraindications, allergies, or previous adverse events or treatment failures with lithium;
* Women who are not currently pregnant and are willing and able to use birth control;
* Are clinically appropriate to treat with lithium.

Exclusion Criteria:

* DSM-IV Axis I Diagnosis: other primary comorbid axis I disorders such as: schizophrenia, schizoaffective disorder, delusional disorder;
* Alcohol or Substance Dependence: meets criteria for dependence within past 3 months;
* Unstable Medial Conditions: Life threatening or unstable medical condition that require active adjustment of medications by medical history; or
* Medical Conditions: concomitant medical condition that would preclude the use of lithium (i.e.: renal failure, head trauma with loss of consciousness, or clinically significant cardiac, renal, hepatic, neoplastic, or cardiovascular disease);
* Concomitant treatment with the following medications (during maintenance Phase): antipsychotics, antidepressants, antianxiety agent with the exception of benzodiazepines, to be used if needed for anxiety or insomnia, not to exceed 10 doses/week, or mood stabilizers with the exception of lithium; and
* Active suicidal or homicidal ideations as elicited in the interviews.
* Stable and doing well on a mood stabilizer other than lithium.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Veterans with bipolar disorder
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2005-10; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Kelsoe, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIMH-sponsored study of the genetics of bipolar disorder — http://www.clinicaltrials.gov/ct2/show/NCT00001174
- See also: National Patient support group for bipolar disorder — http://dbsalliance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with bipolar disorder were recruited through the San Diego VA Mood Clinic
Groups:
- Bipolar Disorder: Veterans with bipolar disorder
  Lithium treatment: Lithium is a standard treatment for bipolar disorder. Patients will be stabilized on lithium monotherapy over a 3 month period, observed for one month, and then followed every 2 months in maintenance phase for 2 years
Period: Overall Study
Arm/Group | Bipolar Disorder
Started | 130
Completed | 110
Not Completed | 20
Not completed — Lost to Follow-up | 20

BASELINE CHARACTERISTICS:
Population: approximately 80 patients were suitable for analysis once lost to followups and other situations where data was not valid.
Arm/Group | Bipolar Disorder
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 116
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 108
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 130

OUTCOME MEASURES:

1. Primary Outcome: Time to Relapse
Description: The primary outcome measure was time to relapse in months following stabilization on lithium.
Time Frame: every 2 months for 2 years
Population: outpatients at VA San Diego Healthcare System
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Bipolar Disorder
Number analyzed (Participants) | 130
months | 24.6 [19.5 to 29.7]

ADVERSE EVENTS:
Time Frame: 10 years
Description: The study is ended.
Groups:
- Bipolar Disorder: Subjects with Bipolar Disorder who are treated with lithium
Arm/Group | Bipolar Disorder
All-Cause Mortality (participants affected / at risk) | 0/130
Serious Adverse Events (participants affected / at risk) | 0/130
Other Adverse Events (participants affected / at risk) | 16/130
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bipolar Disorder (N=130)
weight gain (Metabolism and nutrition disorders) | 16 (16) — weight gain

LIMITATIONS AND CAVEATS:
The study results are limited by small sample size and a dropout rate higher than expected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes